CLINICAL TRIAL: NCT03492996
Title: A Mass Balance Study to Investigate the Absorption, Metabolism, Excretion of LCB01-0371 After a Single Oral LCB01-0371 Dose With a [14C]LCB01-0371- Microtracer Dose in Healthy Male Subjects
Brief Title: A Mass Balance Study of LCB01-0371 After a Single Oral LCB01-0371 Dose With a [14C]LCB01-0371-microtrace
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LigaChem Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCB01-0371-17-1-06
Record Dates: First submitted 2018-04-01; First posted 2018-04-10 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2020-11

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- LCB01-0371 dose with a [14C]-LCB01-0371-tracer (Experimental): A mass balance study to investigate the absorption, metabolism, excretion of LCB01-0371 after a single oral LCB01-0371 dose with a [14C]-LCB01-0371-tracer dose in healthy male subjects
  Interventions: Drug: LCB01-0371 dose with a [14C]-LCB01-0371-tracer dose

INTERVENTIONS:
Drug: LCB01-0371 dose with a [14C]-LCB01-0371-tracer dose — To assess the absorption, metabolism, excretion of LCB01-0371 after a single oral LCB01-0371 dose with a [14C]-LCB01-0371-tracer dose to healthy subjects

SUMMARY:
The primary objectives of the study are:

• To assess the absorption, metabolism, excretion of LCB01-0371 after a single oral LCB01-0371 dose with a [14C]-LCB01-0371-tracer dose to healthy subjects

DETAILED DESCRIPTION:
This is a single-center, open-label, non-randomized, one-sequence, one-period, single arm study in healthy male subjects. A total of 6 subjects will be enrolled in the study, and a minimum of 4 evaluable subjects are considered sufficient. An evaluable subject is defined as a subject who has provided whole blood, plasma, exhalation and excreta samples sufficient for evaluation of the primary objectives. Study subjects will be screened for eligibility to participate in the study within 28 days before dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male adults aged 19 to 45 (inclusive) years
2. Body weight at least 55 kg and calculated Body Mass Index (BMI) ranging from 18.0 to 25.0 kg/m2
3. Subjects who agreed to voluntarily participate in this study and comply with all the protocol requirements by signing informed consent form
4. Subjects who were deemed as eligible subjects by investigators on their physical examination, laboratory findings, and medical examination by interview.
5. Subject who were not to have a history of drug hypersensitivity or allergic reactions related to antibiotics, etc

Exclusion Criteria:

1. Subjects who had a clinically significant disease or a past history of disease
2. Subjects who had a past history of gastrointestinal disease (Crohn's disease, ulcer, acute or chronic pancreatitis, etc.) or surgery (excluding simple appendectomy or hernia surgery) that may have affected to absorption for the study drug.
3. Subjects who had the following laboratory test results at screening; AST, ALT, and total bilirubin ≥ 1.5 times upper limit of normal or CK (Creatine Kinase) > 2.5 times upper limit of normal
4. Subjects who had history of drug abuse or showed a positive result on a drug screening urine test.
5. Subjects who showed a positive result for a serology test (HBsAg, Anti-HCV , HIV Ab, or VDRL), etc.

Ages: 19 Years to 46 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2020-06-21 (Actual); Primary Completion 2020-08-03 (Actual); Study Completion 2020-09-23 (Actual)

PRIMARY OUTCOMES:
Assess the AME of LCB01-0371 | an average of 8 days (+ - 1 D)
  To assess the absorption, metabolism, excretion of LCB01-0371 after a single oral LCB01-0371 dose with a [14C]-LCB01-0371-tracer dose to healthy subjects.
  Blood, urine, feces, and expired air samples will be collected according to the following schedules
  1. Blood: Plasma(20 points), Whole blood(2 points)
  2. Urine : 11 points
  3. Feces : 8 points
  4. Expired air: 14points

CONTACTS AND LOCATIONS:
Overall Officials: Howard Lee, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No